CLINICAL TRIAL: NCT07125677
Title: Comparison of Airway Sealing Pressure Between I-gel® and I-gel Plus® in Elderly Patients Under General Anesthesia
Brief Title: I-gel Plus Comparison Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dongguk University International Hospital (Other)
Responsible Party: Principal Investigator, Hansu Bae, Assistant professor, Dongguk University International Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DUIH 2025-04-012-003
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Airway Management in Elderly Patients Using Supra Glottic Airway Under General Anesthesia
Keywords: I-gel study; SGA study; Elderly patients

STUDY DESIGN:
Intervention Model Description: Prospective crossover design where patients are randomized to receive either I-gel first followed by I-gel plus (Group I) or vice versa (Group P)
Masking Description: No blinding is implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Patients receive I-gel® first, followed by removal and insertion of I-gel plus®.
  Interventions: Device: I-gel first; Behavioral: common
- Group P (Active Comparator): Patients receive I-gel plus® first, followed by removal and insertion of I-gel®.
  Interventions: Device: I-gel plus first; Behavioral: common

INTERVENTIONS:
Device: I-gel first — After general anesthesia, I-gel is inserted first, the maximum sealing pressure is measured, and then it is removed. Subsequently, I-gel plus is inserted, and the same procedure is repeated.
  Arms: Group I
Device: I-gel plus first — After general anesthesia, I-gel plus is inserted first, the maximum sealing pressure is measured, and then it is removed. Subsequently, I-gel is inserted, and the same procedure is repeated.
  Arms: Group P
Behavioral: common — Prior to general anesthesia, as a common baseline procedure for all study arms, the patient's Charlson Comorbidity Index and frailty score are assessed and recorded through patient evaluation (using the Clinical Frailty Scale for the frailty score). Immediately before induction of anesthesia, progressive pressures (100 g, 200 g, 300 g, 400 g, and 500 g) are applied to the patient's thyroid cartilage, and the degree of deviation is measured and documented.

SUMMARY:
This study compares the airway sealing pressure between I-gel® and I-gel plus® in elderly patients (aged 65-85) undergoing general anesthesia. I-gel® is a supraglottic airway device with a non-inflatable cuff, and I-gel plus® is an improved version with a larger gastric drainage channel, enhanced airway tube, and longer cuff tip for better sealing. The study aims to evaluate differences in sealing pressure and other performance metrics in this population, where anatomical changes may affect device efficacy.

DETAILED DESCRIPTION:
Supraglottic airway devices (SGAs) are widely used as alternatives to endotracheal intubation in anesthesiology and emergency medicine. The I-gel® (Intersurgical Ltd., UK) features a non-inflatable cuff for ease of insertion and excellent sealing. The I-gel plus® improves on this with a larger gastric channel, better airway tube, and extended cuff tip to enhance sealing pressure.

Prior studies compared I-gel® to other SGAs like ProSeal or Supreme, showing variable sealing pressures, but direct comparisons between I-gel® and I-gel plus®, especially in elderly patients, are lacking. Elderly patients may experience upper airway anatomical changes affecting SGA performance. Higher sealing pressure is crucial for surgeries with increased intra-abdominal pressure (e.g., laparoscopic or robotic surgery) and can reduce respiratory complications in patients with airway hypersensitivity.

This prospective crossover study will quantitatively assess differences in sealing pressure, fixation stability, and other outcomes. Both devices are approved by the Korean MFDS and will be used within approved indications for academic evaluation of efficacy in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65-85 years with ASA physical status I-III.
* Scheduled for elective surgery under general anesthesia lasting less than 3 hours.

Exclusion Criteria:

* High risk of aspiration (history of gastrectomy, BMI >35 kg/m², gastroesophageal reflux disease, hiatal hernia).
* Poor dental status preventing I-gel fixation.
* Cervical spine instability.
* Anatomical abnormalities in mouth or larynx, or high risk of respiratory complications (asthma, COPD, recent pneumonia).
* Pregnancy.
* Other cases deemed inappropriate by the investigator.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Airway Sealing Pressure | During surgery, immediately after each device insertion
  Comparison of sealing pressure (cm H2O) between I-gel® and I-gel plus®, measured after insertion with fresh gas flow at 3 L/min and valve closed.

SECONDARY OUTCOMES:
Fixation Stability | During surgery
  Assessment of device position maintenance after insertion (device movement yes/no).
Time to Successful Insertion | During surgery
  Time from start of insertion to complete EtCO2 curve appearance (twice).
Ease of Insertion | During surgery
  Graded as 1 (success on first attempt, no resistance), 2 (success on first, with resistance), 3 (success after >1 attempt).
Operator Complications | Post-surgery up to 24 hours
  Incidence of sore throat, laryngospasm, voice hoarseness, dysphagia.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
Data will be managed confidentially and stored for 3 years post-study, then destroyed per privacy laws. No sharing planned.